CLINICAL TRIAL: NCT00966368
Title: A Trial to Test for Bioequivalence Between Two NN1250 Formulations in Healthy Subjects
Brief Title: Comparison of Two NN1250 Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1250-1988; U1111-1122-2992 (Other: WHO); 2011-002949-35 (EudraCT Number); P/44/2010 (Other: EMA (PDCO)); P/96/2011 (Other: EMA (PDCO))
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg E (Experimental)
  Interventions: Drug: insulin degludec
- IDeg M (Experimental)
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — Single dose of NN1250, formulation 1, 0.4U/kg body weight injected subcutaneously (under the skin)
  Arms: IDeg E
Drug: insulin degludec — Single dose of NN1250, formulation 2, 0.4U/kg body weight injected subcutaneously (under the skin)
  Arms: IDeg M

SUMMARY:
This trial was conducted in North America. The aim of this clinical trial was to investigate if two formulations of NN1250 (insulin degludec) have the same level of drug exposure to the body.

ELIGIBILITY:
Inclusion Criteria:

* Considered generally healthy upon completion of medical history, physical examination, vital signs and ECG (electrocardiogram), as judged by the Investigator
* Body mass index 18.0-27.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Area under the Insulin Degludec concentration-time curve from 0 to 120 hours after single dose | From 0 to 120 hours after dosing
Maximum observed Insulin Degludec concentration after single dose | From 0 to 120 hours after dosing

SECONDARY OUTCOMES:
Time to maximum observed Insulin Degludec concentration after single dose | From 0 to 120 hours after dosing
Area under the Insulin Degludec concentration-time curve from 0 to 24 hours after single dose | From 0-24 hours after dosing
Terminal half-life for Insulin Degludec | From 0 to 120 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Clinical Trial Call Center, Chula Vista, California, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com